CLINICAL TRIAL: NCT02415777
Title: Clinical Trial to Evaluate the Efficacy and Safety of 'URSA SOFT CAP. (UDCA-003)' in Fatigue Patients With Liver Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_UDCA003
Record Dates: First submitted 2014-10-08; First posted 2015-04-14 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Ursodeoxycholic Acid; Thiamine; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- udca003 (Experimental): udca003
  Interventions: Drug: Ursodeoxycholic acid, thiamine, riboflavin
- placebo (Placebo Comparator): placebo of udca003
  Interventions: Drug: Ursodeoxycholic acid, thiamine, riboflavin

INTERVENTIONS:
Drug: Ursodeoxycholic acid, thiamine, riboflavin

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of 'URSA SOFT CAP. (UDCA-003)' in fatigue patients with liver dysfunction

ELIGIBILITY:
Inclusion Criteria:

* CIS greater than or equal to 76, HADS less than or equal to 10
* ALT greater than upper limit of normal OR fatty liver on US

Exclusion Criteria:

* Subjects who have diseases that can cause fatigue
* Subjects who are taking medication that can cause fatigue

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rate of subjects whose CIS score has improved under 76 at week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ilsan Paik Hospital, Ilsan, Kyung-gi-do, South Korea

REFERENCES:
- [Derived] Oh B, Choi WS, Park SB, Cho B, Yang YJ, Lee ES, Lee JH. Efficacy and safety of ursodeoxycholic acid composite on fatigued patients with elevated liver function and/or fatty liver: a multi-centre, randomised, double-blinded, placebo-controlled trial. Int J Clin Pract. 2016 Apr;70(4):302-11. doi: 10.1111/ijcp.12790. Epub 2016 Mar 20. PMID 26997458